CLINICAL TRIAL: NCT03900858
Title: Short Course Rifapentine and Isoniazid for the Preventive Treatment of Tuberculosis(SCRIPT-TB)
Acronym: TB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Affiliated Wenling Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director of Division of Infectious Diseases, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017ZX10201302-004
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Silicosis Tuberculosis
Keywords: rifapentine; isoniazid; preventive
MeSH Terms: interventions — rifapentine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isoniazid/ Rifapentine 3 times a week (Experimental): Intervention：Isoniazid/ Rifapentine 3 times a week given by DOT oral Rifapentine (450mg) plus Isoniazid (400mg) for 12 doses
  Interventions: Drug: Isoniazid；Rifapentine
- No Intervention (No Intervention): No preventive treatment Follow up without intervention. Have already done.

INTERVENTIONS:
Drug: Isoniazid；Rifapentine — 1 months (12 doses) of three-weekly rifapentine at a dose of 450mg plus isoniazid at a dose of 400mg given under direct observation
  Other Names: Isoniazid I INH; Rifapentine RPT; 1RPT/INH 1HP
  Arms: Isoniazid/ Rifapentine 3 times a week

SUMMARY:
Tuberculosis (TB) remains the most important infectious disease in the world. Preventive treatment plays an important role in successful control of TB. The investigators' previous study showed a 3-month weekly rifapentine and isoniazid regimen had a high protective efficacy but an unsatisfactory completion rate. Therefore, the investigators suppose that a one-month (12-dose) regimen of rifapentine and isoniazid (1RPT/INH) to be equivalent to a 3-month weekly rifapentine and isoniazid regimen with similar efficacy and higher completion rate. Relevant study is lacking in China where the TB burden is high with the incidence rate of 70/100, 000.

Silicosis is a risk factor of Mycobacterium tuberculosis infection. This is an open-label, non-randomized clinical trial to evaluate the efficacy and safety of the 1RPT/INH to prevent tuberculosis (TB) compared with those who do not receive preventive treatment among silicotic patients.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains the most important infectious disease in the world. Preventive treatment plays an important role in successful control of TB. For preventive therapy, alternative shortened courses such as 1-month daily rifapentine and isoniazid have been evaluated in HIV-infected individuals for its non-inferiority, safety and convenience compared with traditional monotherapy. And the treatment completion rate is higher. The investigators' previous study showed a 3-month weekly rifapentine and isoniazid regimen had a high protective efficacy but an unsatisfactory completion rate. Therefore, the investigators suppose that a one-month (12-dose) regimen of rifapentine and isoniazid (1RPT/INH) to be equivalent to a 3-month weekly rifapentine and isoniazid regimen with similar efficacy and higher completion rate. Relevant study is lacking in China where the TB burden is high with the incidence rate of 70/100, 000.

Silicosis is a risk factor of Mycobacterium tuberculosis infection. This is an open-label, non-randomized clinical trial to evaluate the efficacy and safety of the 1RPT/INH to prevent tuberculosis (TB) compared with those who do not receive preventive treatment among silicotic patients.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with Silica exposure or diagnosed with silicosis;
* Age between 18 to 65 years;
* Willing to provide signed informed consent, or parental consent and participant assent.

Exclusion Criteria:

* Clinical or culture confirmed active TB;
* A history of treatment for > 14 consecutive days with a rifamycin or > 30 consecutive days with INH during the previous 2 years;
* A documented history of a completing an adequate course of treatment for active TB or latent TB infection;
* Allergy to Isoniazid, Rifampin, or Rifapentine;
* Human immunodeficiency virus (HIV) infection;
* History of hepatitis B/C infection or liver cirrhosis;
* Serum Aspartic transaminase (AST) or alanine transaminase (ALT) > 2x upper limit of normal or total bilirubin >2.5 mg/dL;
* Receiving immunosuppressants or biological agents;
* Life expectancy <3 years;
* Mental disorder;
* Participated in other clinical trials in recent three months;
* Other conditions that investigates consider not suitable for participate.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative rate of culture-confirmed or clinically diagnosed TB disease in participants | 3 years
  Cumulative rate of culture-confirmed or clinically diagnosed TB disease in participants

SECONDARY OUTCOMES:
Percentage of participants with drug discontinuation for any reason and due to adverse drug reactions associated with 1RPT/INH | up to 30 days after the last dose of study drug
  Percentage of participants with drug discontinuation for any reason and due to adverse drug reactions associated with 1RPT/INH
Percentage of patients with Grade 3 or 4 drug toxicities and deaths associated with 1RPT/INH | up to 30 days after the last dose of study drug
  Percentage of patients with Grade 3 or 4 drug toxicities and deaths associated with 1RPT/INH
Percentage of participants who complete the treatment regimen | Enrollment up to Month 1 (1RPT/INH)
  Percentage of participants who complete the treatment regimen

CONTACTS AND LOCATIONS:
Overall Officials: Wenhong Zhang, MD，PhD, Principal Investigator — Huashan Hospital of Fudan University，Shanghai，China
Locations (1):
- Wenling No.1 People's Hospital, Zhejiang, Taizhou, Zhejiang, China

REFERENCES:
- [Derived] Ruan QL, Yang QL, Ma CL, Lin MY, Huang XT, Mao YP, Gao JM, Li JJ, Zhang XN, You ZX, Zheng QQ, Ren YF, Liu XF, Shao LY, Zhang WH. Efficacy and safety of a novel short course rifapentine and isoniazid regimen for the preventive treatment of tuberculosis in Chinese silicosis patients: a pilot study (SCRIPT-TB). Emerg Microbes Infect. 2025 Dec;14(1):2502010. doi: 10.1080/22221751.2025.2502010. Epub 2025 May 16. PMID 40326358